CLINICAL TRIAL: NCT05832983
Title: The Effect of Aromatherapy on Situational Anxiety in Adults Receiving Intra-Articular Injections in the Ambulatory Clinic Setting
Brief Title: Aromatherapy and Anxiety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-00170
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Related to Pain Related to an Intraarticular Injection; Pain Related to an Intraarticular Injection
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in the control arm will receive the current standard of nursing care for treating anxiety prior to receiving the intra-articular injection (emotional support, distraction, and/or therapeutic touch as necessary).
- Experimental Group A (Experimental): Participants in Group A will receive a guided meditation prior to receiving the intra-articular injection.
  Interventions: Behavioral: Guided Meditation
- Experimental Group B (Experimental): Participants in Group B will receive an Elequil Aromatab and the same guided meditation delivered to Group A prior to receiving the intra-articular injection.
  Interventions: Behavioral: Guided Meditation; Other: Aromatherapy

INTERVENTIONS:
Behavioral: Guided Meditation — In private exam room, the study registered nurse (RN) will read a prepared two minute guided meditation to patient.
  Arms: Experimental Group A; Experimental Group B
Other: Aromatherapy — In private exam room, study RN will first affix an Elequil Aromatab to patient's clothing on either their upper arm or chest (whichever the patient prefers and/or as clothing allows).
  Other Names: Elequil Aromatab
  Arms: Experimental Group B

SUMMARY:
While intra-articular injections can alleviate pain in orthopedic patients, this can be an anxiety-provoking experience. Adult patients scheduled to receive an injection at the study location will be randomly assigned to one of three groups. The control group (C) will receive the current standard of nursing care. The first experimental group (A) will receive a guided meditation prior to receiving the injection. The second experimental group (B) will receive an Elequil Aromatab and the same guided meditation prior to receiving the injection.

DETAILED DESCRIPTION:
The objective of the study is to measure the difference in anxiety levels of adult orthopedic patients in need of intra-articular injections who receive a guided meditation only prior to their injection, compared to those who receive a guided meditation and an aromatherapy Elequil Aromatab prior to injection, as well as compared with those who receive the usual standard of care

ELIGIBILITY:
Inclusion Criteria:

* Patient has an in-office appointment at the NYU Langone Ambulatory Care-23rd Street location with either the Ortho A & B (primarily those patients who may be seeking knee or hip replacement surgery), Hand, or Primary Sport clinics.
* Patient has an order for an intra-articular injection (as determined by clinic MD) and has consented to receiving that treatment.
* Patient is English speaking.

Exclusion Criteria:

* Patient has a cognitive or physical disability that would interfere with their ability to complete the study's pre and post assessments with RN.
* Patient is found on the pre-injection assessment form to have an intolerance or allergy to lavender, sandalwood, or strong scents in general.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Short-Version Spielberger State-Trait Anxiety Inventory (SSTAI) Score | 10-15 minutes prior to injection, 5 minutes post-injection (Day 1)
  The Short-Version SSTAI is a 10-item self-assessment of anxiety, with 5 items assessing states of anxiety and 5 items assessing traits of anxiety. Each item is scored on a Likert scale ranging from 1 to 4, where (1 = not at all) and (4 = very much so). The total score is the sum of responses and ranges from 10-40; lower scores indicate lower levels of anxiety. A decrease in scores indicates anxiety decreased during the observational period.
Change in Pain Score | 10-15 minutes prior to injection, 5 minutes post-injection (Day 1)
  On a scale of 0 to 10 (0 = no pain, 10 = the worst pain imaginable), participants rank their pain prior to the injection and after the injection. The total score ranges from 0-10, with higher scores indicating greater pain. A decrease in score indicates pain decreased during the observational period.
Change in Blood Pressure | 10-15 minutes prior to injection, 5 minutes post-injection (Day 1)
  Participants will have their blood pressure (systolic/diastolic - mmHg) taken before and after the injection.
Change in Heart Rate | 10-15 minutes prior to injection, 5 minutes post-injection (Day 1)
  Participants will have their heart rate (beats per minute) measured before and after the injection.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Withall, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data to be used for only this study.